CLINICAL TRIAL: NCT01640977
Title: A Prospective Non-current Concurrent Controlled Evaluation of Open and MAS® PLIF for the Treatment of Symptomatic Lumbar Degenerative Conditions
Brief Title: A Prospective Non-concurrent Controlled Evaluation of Open and MAS® PLIF
Status: Completed | Type: Observational
Sponsor: NuVasive (Industry)
Responsible Party: Sponsor
Organization: Globus Medical Inc (Industry)
Other Study IDs: NUVA.P1001
Record Dates: First submitted 2012-07-09; First posted 2012-07-16 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Lumbar Degenerative Disc Disease
Keywords: Open PLIF; MAS PLIF; Lumbar spine
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Open PLIF: The PLIF procedure achieves access to the degenerated disc from the back of the spine, and is performed through a single midline posterior incision that is typically expanded bilaterally past the facet joints to expose bony landmarks for pedicle screw fixation, which are traditionally placed in a trajectory from lateral to medial, requiring a more lateral starting point.
  Interventions: Procedure: Open PLIF (posterior lumbar interbody fusion)
- MAS PLIF: The MAS PLIF technique is a minimally invasive variant of the traditional PLIF procedure. It is similarly performed through a single midline posterior incision but is conducted through a more medialized posterior approach, avoiding the far lateral exposure typical of the traditional PLIF.
  Interventions: Procedure: MAS PLIF

INTERVENTIONS:
Procedure: Open PLIF (posterior lumbar interbody fusion) — The PLIF procedure achieves access to the degenerated disc from the back of the spine.
  Groups: Open PLIF
Procedure: MAS PLIF — The MAS PLIF technique is a minimally invasive variant of the traditional PLIF procedure. It is similarly performed through a single midline posterior incision but is conducted through a more medialized posterior approach.
  Groups: MAS PLIF

SUMMARY:
The study is a prospective non-concurrent controlled observational evaluation of short-term operative results. As such, study sites will capture perioperative (through 6-week postoperative follow-up) case data associated with 10 standard open PLIF (posterior lumbar interbody fusion) procedures. After this open experience, these same sites will capture the corresponding data from 10 subsequent cases where the MAS (Maximum Access Surgery) PLIF variant was performed. The data from both series of cases will be compiled to identify similarities and differences between the techniques.

DETAILED DESCRIPTION:
The objective of this evaluation is to collect and compare short-term factors related to the morbidity of approach using traditional posterior-approach interbody fusion techniques and a less invasive exposure for the same procedure. Perioperative measures and early outcomes will be documented to demonstrate differences in procedural requirements, safety, and early recovery. A total of 100 subjects will be consecutively enrolled in this prospective study from as many as 8 centers. Patients who, in the surgeon investigator's opinion, require instrumented lumbar interbody fusion and have consented to PLIF surgery for their conditions will be included. The following eligibility criteria are designed to identify existing clinic patients for whom study under this protocol is considered appropriate. All subjects must meet the inclusion/exclusion criteria in order to be considered for enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all inclusion criteria to be eligible for enrollment into this observational study:

  1. Indicated for posterior lumbar interbody fusion at one or two contiguous motion segments between L1 and S1;
  2. 18+ years of age at the date of written informed consent;
  3. Able to undergo surgery based on physical exam, medical history and surgeon judgment;
  4. Willing and able to return for post-treatment exams according to the follow-up called for in the protocol;
  5. Signed and dated informed consent form.

     Exclusion Criteria:
* Subjects presenting with any of the following will not be included in this observational study:

  1. Mental or physical condition that would limit the ability to comply with study requirements;
  2. Spine abnormality requiring treatment at more than two levels;
  3. Prior surgery at operative or adjacent level(s);
  4. Involvement in active litigation relating to the spine (worker's compensation claim is allowed if it is not contested);
  5. Significant general illness (e.g., HIV, active metastatic cancer of any type, uncontrolled diabetes, dialysis dependent renal failure, symptomatic liver disease);
  6. Participating in another clinical study that would confound study data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Existing clinic patients
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2012-06; Primary Completion 2014-06 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Complications | 6-weeks
  All complications will be compiled and their incidence and relationship to the product and/or surgical procedure will be tabulated for comparison.

SECONDARY OUTCOMES:
Clinical Outcomes | 6-weeks
  Visual analog scale (for patient self assessment of back/leg pain)
Radiographic Outcomes | 6-weeks
  Radiographic assessment (AP/lateral x-rays)

CONTACTS AND LOCATIONS:
Overall Officials: Kelli Howell, MS, Study Director — NuVasive
Locations (4):
- United States (4):
  - Kuether Brain and Spine, Greensboro, North Carolina
  - Nova Neurosurgical Brain and Spine, Greensboro, North Carolina
  - WellSpan Orthopedics-York, York, Pennsylvania
  - Scott and White Healthcare, Temple, Texas

REFERENCES:
- See also: sponsor website — http://www.nuvasive.com